CLINICAL TRIAL: NCT03851965
Title: A Prospective Observational Study on Assessment of the Soluble Urokinase Plasminogen Activator Receptor in Adult Patients Undergoing Major Non-cardiac Surgery
Brief Title: Assessment of the Soluble Urokinase Plasminogen Activator Receptor in Non-cardiac Surgery (SPARSE)
Acronym: SPARSE
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Athanasios Chalkias, MD, PhD, Asst. Professor of Anesthesiology, University of Thessaly
Other Study IDs: UTHDA-AC01
Record Dates: First submitted 2018-12-17; First posted 2019-02-22 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Surgery--Complications
Keywords: Soluble urokinase plasminogen activator receptor; Major non-cardiac surgery; Outcome; Perioperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Soluble Urokinase Plasminogen Activator Receptor — Preoperative and postoperative determination of the Soluble Urokinase Plasminogen Activator Receptor levels in patients undergoing non-cardiac major surgery.

SUMMARY:
In critically ill patients, the soluble urokinase plasminogen activator receptor (suPAR) level is significantly increased. suPAR is an independent prognostic marker, and the change over time correlates with organ dysfunction. suPAR is elevated and has a prognostic value in patients with systemic inflammatory response syndrome, sepsis/septic shock, burn injuries, and traumatic brain injuries. SPARSE is a prospective observational study aiming to investigate if suPAR measured preoperatively and immediately after surgery can predict the risk of future complications and post-operative mortality in adults following major non-cardiac surgery. Participants will undergo sampling of peripheral venous blood, immediately after arrival to the Operating Room and at the Post-Anesthesia Care Unit, and plasma suPAR levels will be determined. In addition to routine hemodynamic data, sublingual microvascular flow will be measured using noninvasive technology. The primary endpoint will be the presence of complications and/or admission to ICU and/or mortality within the first 60 postoperative days. Target enrollment will be 100 patients.

DETAILED DESCRIPTION:
BACKGROUND

Soluble urokinase plasminogen activator receptor

The biomarker soluble urokinase plasminogen activator receptor (suPAR) is the soluble form of the cell membrane-bound protein urokinase plasminogen activator receptor (uPAR), which is expressed mainly on immune cells, endothelial cells, and smooth muscle cells. uPAR is released during inflammation or immune activation, and therefore the suPAR level reflects the extent of immune activation in the individual. All human beings have a baseline level of suPAR that is individually determined and increases with age. Studies have shown that the suPAR level is associated with morbidity and mortality in a number of acute and chronic diseases and in the general population. The suPAR level is elevated across diseases, and not solely associated with one specific disease. Therefore, suPAR is applicable as a prognostic marker and not as a diagnostic marker. This characteristic may be utilized for risk stratification in unselected patients.

In critically ill patients, the suPAR level is significantly increased. suPAR is an independent prognostic marker, and the change over time correlates with organ dysfunction. suPAR is elevated and has a prognostic value in patients with: SIRS (systemic inflammatory response syndrome), sepsis/septic shock, burn injuries, and traumatic brain injuries. The suPAR level reflects the body's immune response to infections, and the level increases with the severity of the infection. In patients with organ dysfunction, the suPAR value is often a two-digit value. In particular hepatic and renal dysfunction affects the suPAR level.

suPAR in surgery

The suPAR level is elevated in patients with infections, chronic diseases, and cancer compared to healthy individuals. A high suPAR level is associated with increased mortality risk, poor prognosis, postoperative pneumonia, and prosthetic joint infection. suPAR is a well-studied biomarker predicting prognosis, disease severity, and organ dysfunction and is being considered as a marker of the individual's inflammatory status. It has been demonstrated that biomarkers are able to improve triage and are effective in identifying high and low risk patients among acutely admitted patients. Improving the preoperative risk stratification using biomarkers may optimize the patient's clinical outcome.

AIM

SPARSE is a single-center observational study aiming to investigate if suPAR measured preoperatively and immediately after surgery can predict the risk of future complications and post-operative mortality in adults following major non-cardiac surgery.

METHODS

Design

This is a prospective observational study designed in accordance with the declaration of Helsinki. The study will be register at Clinical Trials.gov and will be approved by the Institutional Review Board of the University Hospital of Larisa, under reference number.

Management of Anesthesia and Surgical Procedures

Endotracheal intubation and anesthetic care will be performed according to institutional routine. Intravenous induction of general anaesthesia will include midazolam 0.15-0.35 mg/kg iv over 20-30 seconds, fentanyl 1μg/kg, propofol 1.5-2 mg/kg, ketamine 0.2 mg/kg (intravenous bolus), and rocurnium 0.6 mg/kg. All drugs will be prepared in labelled syringes and induction will be achieved by administration of a predetermined iv bolus dose on the basis of the patient's weight and/or age. Laryngoscopy and intubation will proceed in a standard fashion, while the position of the endotracheal tube will be confirmed by auscultation and capnography/capnometry. The patients will then connected to an automated ventilator (Draeger Primus®; Drägerwerk AG & Co., Lübeck, Germany).

All patients will be ventilated using a lung-protective strategy with tidal volume of 7 mL/kg, positive end-expiratory pressure of 6-8 cmH2O, plateau pressures <30 cmH2O, and recruitment maneuvers repeated every 30 min after tracheal intubation. Maintenance of general anesthesia will include desflurane 1.0 MAC with 40% oxygen and 60% air, while intraoperative dose changes will be left to the anesthesiologist in charge of the patient. Depth of anesthesia (bispectral index-BIS, Covidien, France) will be monitored, with the target ranging between 40 and 60. Normocapnia will be maintained by adjusting the respiratory rate as needed, while normothermia (37ºC) will be maintained throughout the intraoperative period.

Sampling and laboratory measurements

Participants will undergo sampling of peripheral venous blood, immediately after arrival to the OR, and at the Post-Anesthesia Care Unit (PACU). Blood samples drawn from all patients and EDTA plasma will be stored at -80° C until suPAR levels are determined.

Microcirculation flow analysis

In addition to routine hemodynamic data, sublingual microvascular flow will be measured using noninvasive technology. Measurements will be obtained preoperatively (PRE), intraoperatively (INT), and postoperatively after arrival in the PACU (POST). At each time point, the microcirculatory network of the sublingual mucosa will be imaged using sidestream darkfield (SDF+) videomicroscopy which has an increased optical resolution resulting in one pixel recording an area of 0.56 μm2.

Data Collection and Monitoring

Data analysis will be based on predefined data points on a prospective data collection form. The staff will be blinded to measurements until the end of the study and all data are analyzed. Clinical monitoring throughout the study will be performed to maximize protocol adherence, while an independent Data and Safety Monitoring research staff will monitor safety, ethical, and scientific aspects of the study. Data collection will include demographics, anesthesia parameters, C-reactive protein, P-POSSUM score, ACS-NSQIP score, APACHE II, SOFA, and the Charlson Age-Comorbidity Index (Charlson score). A SAS macro based on ICD-10 diagnoses will be used to calculate the Charlson score. Two other simpler models adding predictive value to the ASA classification will be also used; the Surgical Mortality Probability Model and a similar model proposed by Glance and Donati.

ELIGIBILITY:
Inclusion Criteria:

* All operative approaches
* Age ≥ 18 years
* American Society of Anesthesiologists' (ASA) physical status I to IV

Exclusion Criteria:

* Age <18 years
* Any infection within the previous 4 weeks
* Severe liver disease
* Renal replacement therapy pre-operatively
* Previously received transplant
* Allergies
* Inflammatory disorders
* Immune system disorders
* Connective tissue disease
* Administration of opioids during the past week
* Asthma
* Obesity (BMI ≥ 30 kg m-2)
* Mental disability
* Severe psychiatric disease
* Alcohol or other abuse,
* Legal incapacity or limited legal capacity
* Subjects within the exclusion period of another study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who are scheduled to undergo elective major non-cardiac surgery with expected duration ≥2 hours under general anesthesia
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative complications | Within the first 90 postoperative days
  Number of participants with postoperative complications
Number of participants admitted to Intensive Care Unit | Within the first 60 postoperative days
  Number of participants admitted to Intensive Care Unit
Number of deaths | Within the first 60 postoperative days
  Number of deaths

SECONDARY OUTCOMES:
Number of participants with intraoperative complications | During surgery
  Number of participants with desaturation [SpO2 <92% for 3 minutes or more], need for unplanned recruitment maneuvers, hypotension [defined as systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg for 3 minutes or more or need of vasoactive drugs for correction]
Number of participants with need for unplanned vasoactive drugs during surgery | During surgery
  Number of participants with need for vasoactive drugs not planned before and/or continuous infusion during surgery
Number of participants with acute new arrhythmia during sugery | During surgery
  Number of participants with atrial fibrillation, sustained ventricular tachycardia, supraventricular tachycardia, and/or cardiac arrest during surgery
Number of reintubations | At 30 days
  Number of participants being reintubated after extubation
Survival | At 30 days, at 90 days, and at 1 year
  Survival

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Chalkias, MD, PhD, Principal Investigator — University of Thessaly, Faculty of Medicine
Locations (1):
- University Hospital of Larisa, Department of Anesthesiology, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication and for the next 6 months.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Stephens RW, Nielsen HJ, Christensen IJ, Thorlacius-Ussing O, Sorensen S, Dano K, Brunner N. Plasma urokinase receptor levels in patients with colorectal cancer: relationship to prognosis. J Natl Cancer Inst. 1999 May 19;91(10):869-74. doi: 10.1093/jnci/91.10.869. PMID 10340907
- [Background] Svendsen MN, Ytting H, Brunner N, Nielsen HJ, Christensen IJ. Preoperative concentrations of suPAR and MBL proteins are associated with the development of pneumonia after elective surgery for colorectal cancer. Surg Infect (Larchmt). 2006 Oct;7(5):463-71. doi: 10.1089/sur.2006.7.463. PMID 17083312
- [Background] Eugen-Olsen J, Andersen O, Linneberg A, Ladelund S, Hansen TW, Langkilde A, Petersen J, Pielak T, Moller LN, Jeppesen J, Lyngbaek S, Fenger M, Olsen MH, Hildebrandt PR, Borch-Johnsen K, Jorgensen T, Haugaard SB. Circulating soluble urokinase plasminogen activator receptor predicts cancer, cardiovascular disease, diabetes and mortality in the general population. J Intern Med. 2010 Sep;268(3):296-308. doi: 10.1111/j.1365-2796.2010.02252.x. Epub 2010 May 28. PMID 20561148
- [Derived] Laou E, Papagiannakis N, Michou A, Ntalarizou N, Ragias D, Angelopoulou Z, Sessler DI, Chalkias A. Association between mean arterial pressure and sublingual microcirculation during major non-cardiac surgery: Post hoc analysis of a prospective cohort. Microcirculation. 2023 May;30(4):e12804. doi: 10.1111/micc.12804. Epub 2023 Mar 21. PMID 36905347
- [Derived] Chalkias A, Laou E, Kolonia K, Ragias D, Angelopoulou Z, Mitsiouli E, Kallemose T, Smith-Hansen L, Eugen-Olsen J, Arnaoutoglou E. Elevated preoperative suPAR is a strong and independent risk marker for postoperative complications in patients undergoing major noncardiac surgery (SPARSE). Surgery. 2022 Jun;171(6):1619-1625. doi: 10.1016/j.surg.2021.10.012. Epub 2021 Nov 1. PMID 34736789

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT03851965/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT03851965/ICF_001.pdf